CLINICAL TRIAL: NCT07355374
Title: Patients With Esophageal Carcinoma Undergoing Minimally Invasive Ivor Lewis Esophagectomy With or Without Intraoperative Endoscopic Pylorus Balloon Dilation: A Randomized Controlled Trial Investigating the Benefits of Intraoperative Endoscopic Pylorus Dilation
Brief Title: Balloon Dilation in Patients Undergoing Minimally Invasive Ivor Lewis Esophagectomy and Its Effect on Reducing DGCE
Acronym: WIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Digestive Health Care Center Basel, Clarunis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-01877
Record Dates: First submitted 2025-11-14; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Delayed Gastric Conduit Emtpying (DGCE); Minimally-invasive Esophagectomy
Keywords: Balloon dilatation; intraoperatively; ivor lewis Esophagectomy; Delayed gastric conduit emtpying (DGCE)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dilation Group (Active Comparator): Intervention group; patients receive additional dilation of the pylorus
  Interventions: Procedure: endoscopic plyoric balloon dilatation performed by experienced gastroenterologists
- Control (No Intervention): In this group patients will undergo standard care without additional intervention

INTERVENTIONS:
Procedure: endoscopic plyoric balloon dilatation performed by experienced gastroenterologists — Standard endoscopic plyoric balloon dilatation performed by experienced gastroenterologists as it would be performed to treat DGCE
  Arms: Dilation Group

SUMMARY:
Background:

Esophageal carcinoma ranks among the most common and lethal cancers worldwide. Minimally invasive esophagectomy is the standard curative treatment, but postoperative delayed gastric conduit emptying (DGCE) remains a major complication, occurring in up to 40% of patients. DGCE prolongs recovery, increases morbidity, and raises healthcare costs. Mechanical stretching of the pylorus has shown potential to reduce DGCE in retrospective studies, but evidence from randomized controlled trials in the context of minimally invasive surgery is lacking.

Objective:

The WIDE Trial aims to evaluate whether intraoperative endoscopic balloon dilation of the pylorus during minimally invasive Ivor-Lewis esophagectomy can reduce the incidence of early postoperative DGCE, improve recovery, and enhance quality of life.

Design:

This is a prospective, single-center, double-blinded, superiority randomized controlled trial conducted at Clarunis University Digestive Health Care Center, Basel. A total of 116 patients with histologically confirmed esophageal carcinoma undergoing minimally invasive esophagectomy with curative intent will be randomized 1:1 into an intervention group and a control group.

Intervention group: Intraoperative endoscopic balloon dilatation of the pylorus to 30 mm before gastric conduit formation.

Control group: Standard minimally invasive Ivor Lewis esophagectomy without dilatation.

Endpoints:

Primary endpoint: Incidence of early DGCE within 14 days postoperatively, defined by radiological and clinical criteria (gastric tube output >500 mL on day ≥5 or >100% increase in gastric tube width on X-ray).

Secondary endpoints: Late DGCE incidence (after >14 days), anastomotic leak rate, overall postoperative complications (Clavien-Dindo classification), hospital stay, time to first bowel movement, time to solid food intake, and postoperative quality of life (EORTC QLQ-OES18).

Methods and Follow-up:

Baseline data are collected preoperatively; postoperative outcomes are assessed at days 5, 10, and 3 months. Ward physicians and radiologists assessing outcomes are blinded to group assignment. At three months, all patients undergo follow-up including symptom questionnaires, radiological passage study, and QoL assessment.

Statistics:

Power analysis (α = 0.05, β = 0.20) based on prior studies suggests that 52 patients per group are needed to detect a reduction in DGCE incidence from 48% to 22%. Accounting for 10% attrition, 116 total patients will be enrolled. Analyses will follow the intention-to-treat principle using chi-square, t-tests/Mann-Whitney U tests, and multivariable logistic regression to adjust for confounders.

Risk-Benefit Assessment:

The intervention poses minimal additional risk, as balloon dilatation is an established and safe endoscopic procedure, adding approximately 20-30 minutes to surgical time. Possible complications such as perforation or bleeding are rare and manageable intraoperatively. Potential benefits include reduced DGCE incidence, shorter hospitalization, lower complication rates, and improved patient quality of life.

Ethics and Data Protection:

The study complies with the Declaration of Helsinki, ICH-GCP, and Swiss ClinO regulations (risk category A). All participants provide written informed consent. Patient data are pseudonymized and securely stored in a REDCap database.

Timeline:

Start of recruitment: December 2025

End of recruitment / last surgery: June 2028

Follow-up: 3 months per patient postoperatively

Expected Impact:

If intraoperative endoscopic pylorus dilatation proves effective, it could become a new standard adjunct procedure in minimally invasive esophagectomy, reducing DGCE-related morbidity and improving recovery and cost-efficiency in esophageal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Histologically confirmed esophageal cancer
* Planned surgical resection in curative intent as a minimally invasive Ivor Lewis procedure
* Provided informed consent

Exclusion Criteria:

* Prior esophageal or gastric resection
* Non-curative intent of surgery
* ASA Score V
* Patients lacking capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Early Delayed Gastric Conduit Emptying (DGCE) on day 5 and 10 | On postoperative day 5 and day 10 after the Intervention and the day of the esophagectomy.
  Early DGCE is defined as:
  >500ml output of the nasogastric tube OR >100% increased gastric tube width on frontal X-Ray. If either one of the mentioned parameters is fullfilled DGCE is present. The Incidence of DGCE is our primary outcome and it is defined by one of the above mentioned criteria.

SECONDARY OUTCOMES:
Incidence of Late DGCE | Data will be collected 3 months after the intervention
  After 3 months postoperatively (after the Intervention) patients are asked to fill out the DGCE symptom questionnaire and a radiological passage will be performed after 3 months to assess the passage of the contrast agent trough the GI-System.
  Late DGCE is defined as: quite a bit or very much of at least 2 of 5 symptoms in the DGCE Quesitonniare and a verdict by the radiologist "delayed contrast passage".
Demographics | Demographic data will be collected prior to the Intervention on day X before the surgery in the surgical consultation, where patients provide the informed consent to participate in the study.
  Demographical data: age, gender are collected for comparison of the results and potential confounders.
Weight | Baseline Day of the Intervention (Before the Intervention)
  Body weight in kilograms at the time of the preoperative anesthesia consultation will be recorded
Perioperative parameters | Data will be collected 3 months after the intervention
  Data concerning hospital and ICU stay (in days after Intervention) are collected for later analysis.
Past medical history | Demographic data and past medical history will be collected prior to the Intervention on day X before the surgery in the surgical consultation, where patients provide the informed consent to participate in the study.
  Past medical history are noted for comparison of the results and potential confounders.
Rate of anastomotic leak | Data will be collected 3 months after the intervention
  The anastomotic leak rate (diagnosed by endoscopy) will be recorded
Complication rate | Data will be collected 3 months after the intervention
  All patients' complication rates will be recorded for comparison
First bowel movement | At discharge (assessed up to 5 days)
  Time (in days) till first bowel movement after the operation is recorded
Postoperative quality of life | Data is collected 3 months after the intervention
  Postoperative quality of life will be assessed using the EORTC QLQ-OES18 questionnaire. Between 18 and 72 points can be reached. Higher scores indicate stronger symptoms and therefore lower quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Beat Müller, Prof., Study Director — Clarunis, University digestive health care centre basel
Locations (1):
- Clarunis University Digestive Health Care Center Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The data will be shared in an anonymized manner to protect participant privacy and prevent data breaches. Data sharing without pseudonymization is not permitted under Swiss ethical and regulatory requirements.

REFERENCES:
- [Background] Boshier PR, Adam ME, Doran S, Muthuswamy K, Hanna GB. Effects of intraoperative pyloric stretch procedure on outcomes after esophagectomy. Dis Esophagus. 2018 Oct 1;31(10). doi: 10.1093/dote/doy038. PMID 29846516
- [Background] Nienhuser H, Heger P, Crnovrsanin N, Schaible A, Sisic L, Fuchs HF, Berlth F, Grimminger PP, Nickel F, Billeter AT, Probst P, Muller-Stich BP, Schmidt T. Mechanical stretching and chemical pyloroplasty to prevent delayed gastric emptying after esophageal cancer resection-a meta-analysis and review of the literature. Dis Esophagus. 2022 Jul 12;35(7):doac007. doi: 10.1093/dote/doac007. PMID 35178557
- [Background] Konradsson M, van Berge Henegouwen MI, Bruns C, Chaudry MA, Cheong E, Cuesta MA, Darling GE, Gisbertz SS, Griffin SM, Gutschow CA, van Hillegersberg R, Hofstetter W, Holscher AH, Kitagawa Y, van Lanschot JJB, Lindblad M, Ferri LE, Low DE, Luyer MDP, Ndegwa N, Mercer S, Moorthy K, Morse CR, Nafteux P, Nieuwehuijzen GAP, Pattyn P, Rosman C, Ruurda JP, Rasanen J, Schneider PM, Schroder W, Sgromo B, Van Veer H, Wijnhoven BPL, Nilsson M. Diagnostic criteria and symptom grading for delayed gastric conduit emptying after esophagectomy for cancer: international expert consensus based on a modified Delphi process. Dis Esophagus. 2020 Apr 15;33(4):doz074. doi: 10.1093/dote/doz074. PMID 31608938

DOCUMENTS (1):
  • Study Protocol (2025-12-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT07355374/Prot_000.pdf